CLINICAL TRIAL: NCT02901158
Title: Esophageal Manometry in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Lundin, Professor, Sahlgrenska University Hospital
Other Study IDs: LUA-74203
Record Dates: First submitted 2016-09-09; First posted 2016-09-15 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Acute Respiratory Failure
Keywords: esophageal pressure; chest wall elastance; lung elastance; transpulmonary pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critical care patients: Mechanically ventilated patients in the critical care unit
- OR-patients: Mechanically ventilated patients in the operating room

SUMMARY:
Esophageal pressure measurements are used in to determine chest wall elastance and calculate lung elastance and transpulmonary pressure in mechanically ventilated patients. A dedicated esophageal balloon catheter is then placed in the esophagus to measure tidal variations in esophageal pressure.

In this study high resolution solid-state manometry technique was used to provide detailed and continuous measurements of esophageal pressures in the different parts of the esophagus. Measurements were performed during ongoing mechanical ventilation at different levels of endexpiratory pressure.

DETAILED DESCRIPTION:
Esophageal pressure measurements are used in to determine chest wall elastance and calculate lung elastance and transpulmonary pressure in mechanically ventilated patients. A dedicated esophageal balloon catheter is then placed in the esophagus to measure tidal variations in esophageal pressure.

In this study high resolution solid-state manometry technique was instead used to provide detailed and continuous measurements of esophageal pressures in the different parts of the esophagus. The manometry catheter has 36 circumferential sensors at 1 cm intervals. Each sensor has 12 pressure-sensitive segments that add to the signal at that location. Measurements were performed during ongoing mechanical ventilation at different levels of endexpiratory pressure. Possible differences in tidal variations in esophageal pressure in different parts of the esophagus were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the critical care unit receiving mechanical ventilation or Patients anesthetized and undergoing surgery

Exclusion Criteria:

* Patients with a contraindication to insert a catheter in the esophagus for instance due to an operation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients in the critical care unit and in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Esophageal pressure measurements in mechanically ventilated patients | Within one hour
  Esophageal pressure was measured in mechanically ventilated patients in the critical care unit and in the operating room.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lundin, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persson P, Ahlstrand R, Gudmundsson M, de Leon A, Lundin S. Detailed measurements of oesophageal pressure during mechanical ventilation with an advanced high-resolution manometry catheter. Crit Care. 2019 Jun 13;23(1):217. doi: 10.1186/s13054-019-2484-8. PMID 31196203